CLINICAL TRIAL: NCT05865938
Title: PASCAL vs. MitralClip for Mitral Valve Transchatheter Edge-to-Edge Repair: A Prospective, Single-center, Open-label Study
Brief Title: PASCAL vs. MitralClip for Mitral Valve Transchatheter Edge-to-Edge Repair
Status: Completed | Type: Observational
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Sponsor
Other Study IDs: PASCAL vs. MitralClip
Record Dates: First submitted 2023-05-08; First posted 2023-05-19 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Mitral Regurgitation; Functional Mitral Regurgitation; Degenerative Mitral Valve Regurgitation
Keywords: Mitral Regurgitation; Functional Mitral Regurgitation; Degenerative Mitral Valve Regurgitation; M-TEER; TEER
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PASCAL-Group: M-TEER using MitraClip
  Interventions: Device: PASCAL vs. MitraClip
- MitraClip-Group: M-TEER using PASCAL
  Interventions: Device: PASCAL vs. MitraClip

INTERVENTIONS:
Device: PASCAL vs. MitraClip — transcatheter mitral valve repair of the mitral valve (M-TEER) using the Edwards PASCAL Transcatheter Valve Repair System or the Abbott MitraClip in patients with severe and symptomatic degenerative or functional mitral regurgitation (FMR).
  The type of device system used was not randomized but was determined by the operational structuring of the mitral valve program such that patients were scheduled for the next available implantation date with weekly alternating time slots for MitraClip device and PASCAL device.

SUMMARY:
Comparsion of the current two available TEER systems, the MitraClip with the PASCAL repair system in terms of their effectiveness and safety in patients with degenerative mitral regurgitation (DMR) and in patients with functional regurgitation (FMR), who were referred for an interventional therapy by the heart team due to a high surgical risk profile.

DETAILED DESCRIPTION:
A prospective single-center, open-label study to evaluate the safety and effectiveness of transcatheter mitral valve repair of the mitral valve (M-TEER) using the Edwards PASCAL Transcatheter Valve Repair System compared to using the Abbott MitraClip in patients with severe and symptomatic degenerative or functional mitral regurgitation (FMR). The type of device system used was not randomized but was determined by the operational structuring of our mitral valve program such that patients were scheduled for the next available implantation date with weekly alternating time slots for MitraClip device and PASCAL device. Treating physicians had no influence on scheduling or system selection.

Follow-up examinations will be performed one month and one year after the procedure with assessment of echocardiographic and functional status based on the New York Heart Association (NYHA) grade. Patient characteristics, baseline data, and data related to the procedure were assessed using a registry, medical records and the procedure protocols.

This study is a subproject of the MitraClip® Registry (NCT02033811)

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Severe Mitral Regurgitation (3+ to 4+)
* Symptom status: NYHA functional class ≥ II
* Patients with FMR or DMR, who were referred for M-TEER by the heart team decision due to a high

Exclusion Criteria:

* Life expectancy < 1 year
* Anatomy of the mitral valve that may not be suitable for the MitraClip or PASCAL device
* Contraindication for transoesophageal echocardiography
* Active endocarditis
* Pregnant or planning pregnancy within next 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe symptomatic mitral regurgitation.
Sampling Method: Probability Sample
Enrollment: 214 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Procedural success | one month after implantation
  as defined by the Mitral Valve Academy Research Consortium (MVARC)
Composite endpoint of all-cause death and heart failure hospitalization | one year after implantation

SECONDARY OUTCOMES:
Grade of Mitral Regurgitation | one month and one year after implantation
  measured by echocardiography
Functional status | one month and one year after implantation
  according to New York Heart Association (NYHA) functional class

CONTACTS AND LOCATIONS:
Overall Officials: Malte Kelm, Prof., Study Chair — Clinic for Cardiology, Pneumology and Angiology at University Hospital Düsseldorf; Patrick Horn, MD, Principal Investigator — Clinic for Cardiology, Pneumology and Angiology at University Hospital Düsseldorf; Jafer Haschemi, MD, Principal Investigator — Clinic for Cardiology, Pneumology and Angiology at University Hospital Düsseldorf
Locations (1):
- Division of Cardiology, Pulmonary Disease and Vascular Medicine, Düsseldorf, Germany

IPD SHARING:
Plan to Share IPD: No